CLINICAL TRIAL: NCT02415738
Title: Changes in Cerebral Oxygenation During the Prone Position in Patients With Acute Respiratory Distress Syndrome
Acronym: OXYDV
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Bretagne Atlantique (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-005-YF
Record Dates: First submitted 2015-04-09; First posted 2015-04-14 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: ARDS; Prone Positioning
Keywords: Near infrared spectroscopy; Cerebral oxygenation; Acute respiratory distress syndrom; Prone positioning
MeSH Terms: interventions — Prone Position

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Prone positioning

SUMMARY:
Hypoxemia may be refractory to protective ventilation during the acute respiratory distress syndrome (ARDS), justifying the use of other therapies that improved oxygenation and decreased mortality, including prone position (PP).

During ARDS, the majority of patients are responders to PP with increased PaO2 due to homogenization of the ventilation-perfusion ratio. Despite changes in intra-thoracic and intra-abdominal pressure, hemodynamic parameters are not changed.

Besides the fact that the PP improves systemic oxygenation is it the same on cerebral oxygenation? No study has investigated the cerebral oxygenation during PP in patients with ARDS. The cerebral oxygenation may be altered due to the position of the patient and high levels of positive end-expiratory pressure. This decrease oxygenation may be responsible for cognitive impairment when patients awake.

NIRS (Near Infrared Spectroscopy) is a noninvasive tool, capable of delivering information on cerebral oxidative metabolism and its hemodynamic status. It can be used routinely for the management of resuscitation in Intensive Care Unit (ICU) patients. This study is to investigate cerebral oxygenation during prone position in the investigators' patients of ICU.

DETAILED DESCRIPTION:
Primary objectiv Is there a correlation between rSO2 and SpO2 during prone position in patients with ARDS?

Inclusion criteria

Patient with moderate and severe ARDS from 12h, defined by:

* Acute onset of respiratory failure
* Parenchymal opacities Bilateral not fully explained by pleural effusion, nodules, masses or atelectasis
* Unexplained cardiac or vascular insufficiency filling respiratory distress
* PaO2 / FiO2 ≤ 200 with FiO2> 60% and PEEP ≥ 5cmH2O
* Need for invasive mechanical ventilation
* Hemoglobin> 8 g / dL
* Ramsay score 6 sedated with midazolam and Sufentanyl and neuromuscular blockade by Atracurium.

Exclusion criteria

* Participation in another study requiring specific management of ARDS;
* Against-indication for prone position:

  * Burns or wounds in the face, chest and abdominal wall
  * Recent thoraco-abdominal surgical incision
  * Spinal instability, pelvic fracture
  * State of uncontrolled shock
  * intracranial hypertension
* Alteration of the NIRS signal:

  * Brain damage: extra-dural hematoma, subdural hematoma, pneumocephalus, ischemic stroke, subarachnoid hemorrhage, intracerebral expansive process
  * Skin lesions at the electrodes
  * Jaundice bilirubin
  * ECMO
  * Pregnant or breastfeeding women
  * Age less than 18 years
  * Opposition patient, a family member, person of trust or the legal representative for participation in the study.

ELIGIBILITY:
Inclusion Criteria:

Patient with moderate and severe ARDS from 12h, defined by:

* Acute onset of respiratory failure
* Parenchymal opacities Bilateral not fully explained by pleural effusion, nodules, masses or atelectasis
* Unexplained cardiac or vascular insufficiency filling respiratory distress
* PaO2 / FiO2 ≤ 200 with FiO2> 60% and PEEP ≥ 5cmH2O
* Need for invasive mechanical ventilation
* Hemoglobin> 8 g / dL
* Ramsay score 6 sedated with midazolam and Sufentanyl and neuromuscular blockade by Atracurium.

Exclusion Criteria:

* Participation in another study requiring specific management of ARDS;
* Against-indication for prone position:

  * Burns or wounds in the face, chest and abdominal wall
  * Recent thoraco-abdominal surgical incision
  * Spinal instability, pelvic fracture
  * State of uncontrolled shock
  * intracranial hypertension
* Alteration of the NIRS signal:

  * Brain damage: extra-dural hematoma, subdural hematoma, pneumocephalus, ischemic stroke, subarachnoid hemorrhage, intracerebral expansive process
  * Skin lesions at the electrodes
  * Jaundice bilirubin
  * ECMO
  * Pregnant or breastfeeding women
  * Age less than 18 years
  * Opposition patient, a family member, person of trust or the legal representative for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ARDS
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2015-04; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Brain oxygenation | 18 hours

CONTACTS AND LOCATIONS:
Locations (1):
- CHBA, Vannes, France